CLINICAL TRIAL: NCT07367126
Title: Presence of Neuropathic Pain in Knee Osteoarthritis: Relationship Between Pain Severity and Functional Status
Brief Title: Neuropathic Pain in Knee Osteoarthritis: Pain Severity and Functional Status
Status: Recruiting | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Eser Kalaoglu, Principal Investigator, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Other Study IDs: İstPRMTRH-EK6
Record Dates: First submitted 2026-01-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthristis
Keywords: Pain Intensity; Functional Status; Neuropathic Pain; Knee Osteoarthritis
MeSH Terms: conditions — Pain; Neuralgia; Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 (Case): Patients with Knee OA and Neuropathic Pain (DN4 score ≥ 4)
  Interventions: Other: Clinical and Functional Assessment
- Group 2 (Control): Patients with Knee OA without Neuropathic Pain (DN4 score < 4)
  Interventions: Other: Clinical and Functional Assessment

INTERVENTIONS:
Other: Clinical and Functional Assessment — All participants will undergo a one-time, cross-sectional clinical assessment. Comprehensive demographic and clinical data, including age, body mass index (BMI), educational level, occupation, and marital status, will be recorded for each participant. Pain intensity will be measured using a 10-cm Visual Analog Scale (VAS). Functional status and symptoms related to knee osteoarthritis will be evaluated using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and the Knee Injury and Osteoarthritis Outcome Score-Physical Function Short Form (KOOS-PS). To ensure consistency and minimize measurement error, all anthropometric measurements, specifically weight and height, will be performed by the same researcher.

SUMMARY:
Osteoarthritis (OA) is a degenerative joint disease characterized by structural changes such as cartilage loss and osteophyte formation, leading to functional limitations and disability. Pain in knee OA involves a complex pathophysiological structure including both nociceptive and neuropathic mechanisms. Identifying the neuropathic pain component is clinically significant for improving quality of life and functional recovery. This cross-sectional controlled clinical study aims to determine the prevalence of neuropathic pain in patients with knee OA and evaluate its impact on pain severity and functional status. Patients will be categorized based on the Douleur Neuropathique 4 (DN4) questionnaire and assessed using various pain and functional scales.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a degenerative joint disease characterized by structural alterations, including focal cartilage loss, osteophyte formation, subchondral sclerosis, and synovitis. Given the growing elderly population, the prevalence of OA is rising, frequently leading to significant functional limitations and disability. Pain, the most prominent symptom of OA, serves as a critical measure for monitoring disease activity and treatment efficacy.

Recent evidence suggests that OA-related pain involves a complex pathophysiological structure, incorporating both nociceptive and neuropathic mechanisms. Studies indicate that approximately 19-37% of patients with knee OA exhibit symptoms consistent with neuropathic pain. Identifying this neuropathic component is clinically essential, as it may respond differently to conventional analgesics; thus, recognizing it is vital for optimizing functional recovery and quality of life.

This cross-sectional controlled clinical trial aims to determine the prevalence of neuropathic pain in patients with knee OA and evaluate its impact on pain severity and functional status. Participants diagnosed with knee OA according to the American College of Rheumatology (ACR) criteria will be recruited and categorized into two groups based on a Douleur Neuropathique 4 (DN4) questionnaire score threshold of 4/10.

For all participants, comprehensive demographic and clinical data, including age, body mass index (BMI), educational level, occupation, and marital status, will be recorded. To ensure consistency and minimize measurement error, all anthropometric assessments will be performed by a single researcher. The following standardized assessment tools will be administered to all participants: Visual Analog Scale (VAS), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), and Knee Injury and Osteoarthritis Outcome Score-Physical Function Short Form (KOOS-PS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Knee OA according to ACR criteria.
* Knee pain for more than 3 months.
* Voluntary participation.

Exclusion Criteria:

* History of surgical intervention in the affected knee.
* History of trauma to the affected knee within the last 6 months.
* History of intra-articular injections (e.g., corticosteroids, hyaluronic acid, PRP) or physical therapy involving the affected knee within the last 6 months.
* Presence of severe psychiatric disorders such as severe depression, anxiety disorder, or psychosis.
* Diagnosis of central nervous system diseases, including Parkinson's disease or multiple sclerosis.
* Diagnosis of inflammatory arthritis, such as Rheumatoid Arthritis or Ankylosing Spondylitis.
* Severe cognitive impairment.
* Chronic decompensated cardiac, renal, or hepatic failure.
* Severe psychiatric, neurological, or kognitive disorders.

Decompensated cardiac, renal, or hepatic failure.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source population for this cross-sectional controlled study is the adult patient population diagnosed with knee osteoarthritis (OA) according to the American College of Rheumatology (ACR) criteria, recruited from the Physical Medicine and Rehabilitation outpatient clinic at Istanbul Physical Therapy and Rehabilitation Training and Research Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2025-12-20 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | at baseline assessment
  Pain intensity was assessed using a 10 cm scale, where one end represents "no pain" and the other represents "most severe pain." Patients were asked to rate their pain on a scale from 0 (no pain) to 10 (most severe pain)
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | at baseline assessment
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) consists of subscales evaluating pain (5 items), stiffness (2 items), and physical function (17 items). Using a 5-point Likert scale, scores range from 0 (representing the best status/no pain) to 96 (representing the worst status/extreme pain).

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score - Physical Function Short Form (KOOS-PS) | at baseline assessment
  Knee Injury and Osteoarthritis Outcome Score - Physical Function Short Form (KOOS-PS) is used to evaluate physical functional limitations associated with knee osteoarthritis. It consists of seven items scored on a 5-point Likert scale. Raw scores are converted to a 0-100 scale, where higher scores indicate better physical function.

CONTACTS AND LOCATIONS:
Overall Officials: Eser Kalaoglu, M.D., Principal Investigator — Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Locations (1):
- Istanbul Physical Medicine and Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including all demographic, clinical, and primary/secondary outcome measures will be shared with qualified researchers. The sharing period will commence 6 months after article publication and conclude 1 year thereafter. Data access requests must be accompanied by a methodologically sound proposal and will be granted upon the corresponding author's approval and the execution of a Data Use Agreement (DUA) to strictly ensure confidentiality and adherence to ethical guidelines.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months and ending 1 year following article publication
Access Criteria: Qualified researchers who present a methodologically robust proposal aimed at fulfilling the objectives of the approved project

REFERENCES:
- [Result] Ohtori S, Orita S, Yamashita M, Ishikawa T, Ito T, Shigemura T, Nishiyama H, Konno S, Ohta H, Takaso M, Inoue G, Eguchi Y, Ochiai N, Kishida S, Kuniyoshi K, Aoki Y, Arai G, Miyagi M, Kamoda H, Suzkuki M, Nakamura J, Furuya T, Kubota G, Sakuma Y, Oikawa Y, Suzuki M, Sasho T, Nakagawa K, Toyone T, Takahashi K. Existence of a neuropathic pain component in patients with osteoarthritis of the knee. Yonsei Med J. 2012 Jul 1;53(4):801-5. doi: 10.3349/ymj.2012.53.4.801. PMID 22665349
- [Result] Hochman JR, Davis AM, Elkayam J, Gagliese L, Hawker GA. Neuropathic pain symptoms on the modified painDETECT correlate with signs of central sensitization in knee osteoarthritis. Osteoarthritis Cartilage. 2013 Sep;21(9):1236-42. doi: 10.1016/j.joca.2013.06.023. PMID 23973136
- [Result] Davis MP. What is new in neuropathic pain? Support Care Cancer. 2007 Apr;15(4):363-72. doi: 10.1007/s00520-006-0156-0. Epub 2006 Nov 28. PMID 17131133
- [Result] Treede RD, Jensen TS, Campbell JN, Cruccu G, Dostrovsky JO, Griffin JW, Hansson P, Hughes R, Nurmikko T, Serra J. Neuropathic pain: redefinition and a grading system for clinical and research purposes. Neurology. 2008 Apr 29;70(18):1630-5. doi: 10.1212/01.wnl.0000282763.29778.59. Epub 2007 Nov 14. PMID 18003941
- [Result] Perrot S. Osteoarthritis pain. Best Pract Res Clin Rheumatol. 2015 Feb;29(1):90-7. doi: 10.1016/j.berh.2015.04.017. Epub 2015 May 16. PMID 26267003
- [Result] Pereira D, Peleteiro B, Araujo J, Branco J, Santos RA, Ramos E. The effect of osteoarthritis definition on prevalence and incidence estimates: a systematic review. Osteoarthritis Cartilage. 2011 Nov;19(11):1270-85. doi: 10.1016/j.joca.2011.08.009. Epub 2011 Aug 24. PMID 21907813